CLINICAL TRIAL: NCT05026112
Title: The Arrhythmogenic Potential of Midwall Septal Fibrosis in Dilated Cardiomyopathy: a Combined ECGI and CMR Investigative Study
Brief Title: The Arrhythmogenic Potential of Midwall Septal Fibrosis in Dilated Cardiomyopathy
Acronym: DCM-MSF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 143656
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample collection - for storage of DNA, RNA, small molecule analysis, and blood cells for human induced pluripotent cells.
  Urine sample collection for small molecule analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- DCM with MSF (MSF+): Patients with dilated cardiomyopathy and midwall septal fibrosis identified in a previous cardiac MRI scan
  Interventions: Diagnostic Test: ECG-Imaging; Diagnostic Test: Cardiac MRI scan
- DCM without MSF (MSF-): Patients with dilated cardiomyopathy but without midwall septal fibrosis on previous cardiac MRI scan
  Interventions: Diagnostic Test: ECG-Imaging; Diagnostic Test: Cardiac MRI scan
- Control - MSF+: Control healthy volunteers (HV) to the MSF+ cohort
  Interventions: Diagnostic Test: ECG-Imaging; Diagnostic Test: Cardiac MRI scan
- Control - MSF-: Control healthy volunteers (HV) to the MSF- cohort
  Interventions: Diagnostic Test: ECG-Imaging; Diagnostic Test: Cardiac MRI scan

INTERVENTIONS:
Diagnostic Test: ECG-Imaging — ECG imaging acquisition
Diagnostic Test: Cardiac MRI scan — Cardiac MRI scan

SUMMARY:
Midwall septal fibrosis (MSF) is a common structural abnormality in non-ischaemic dilated cardiomyopathy (DCM). Its presence is believed to increase the risk of malignant ventricular arrhythmias (VA), but the mechanism of arrhythmogenicity is not known. This is particularly relevant in DCM patients with MSF and mid-range left ventricular ejection fraction (LVEF) as they do not currently fulfil criteria for a primary prevention implantable cardioverter-defibrillator (ICD) insertion.

Access to the epicardium for electrical measurements of the heart can enhance the understanding of arrhythmogenicity in DCM, however direct epicardial access is invasive. Instead, the investigators will non-invasively combine high resolution 256-lead ECG imaging (ECGI) and latest generation cardiovascular magnetic resonance (CMR) to study the hearts of 60 DCM patients with and without MSF regardless of LVEF, and 60 matched healthy volunteers. The investigators recently invented the re-usable and CMR-safe SMART-ECGI vest technology for this purpose. Using supercomputers, the investigators will fuse the collected ECGI/CMR data and run electromechanical simulations of whole-heart activation to non-invasively measure each participant's personalised risk of malignant VA induction.

By panoramically mapping the DCM heart in a single beat, the investigators aim to elucidate how MSF perturbs the cardiac activation front and how this could lead to life-threatening VA. This has the potential to change the method by which cardiologists risk stratify patients with DCM.

ELIGIBILITY:
Inclusion Criteria:

* Adults with dilated cardiomyopathy
* With and without midwall septal fibrosis on previous CMR

Exclusion Criteria:

* Needle-phobic patients that would preclude cannulation for contrast injection and blood taking
* anyone unwilling to consent
* anyone with a conventional contraindication for CMR
* anyone with any condition precluding full participation in the study such as DCM patients with infarct-pattern LGE, or subepicardial LGE or non-septal midwall fibrosis (participants with small volume right ventricular insertion point LGE will not be excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with dilated cardiomyopathy, with and without midwall septal fibrosis on previous CMR
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The relationship between the electrical and structural substrate in DCM | 2 years
  The investigators will describe the relationship between the electrical and structural substrate in DCM across the spectrum of left ventricular dysfunction.

SECONDARY OUTCOMES:
Comparison of epicardial activation and conduction patterns via ECGI | 2 years
  The investigators will compare participants with MSF+DCM, MSF-DCM and controls in terms of epicardial activation and conduction patterns (via ECGI).
Comparison of MSF+DCM, MSF-DCM and controls' electromechanical function of the heart via modelling | 2 years
  The investigators will compare MSF+DCM, MSF-DCM and controls in terms of Electromechanical function of the heart (via 4-dimensional computational models)
Personalised simulation of risk of malignant ventricular arrhythmia | 2 years
  Applying and exploring simulation methodology to establish predictions for likely propensity to malignant VA (personalised simulations of risk) between MSF+DCM, MSF-DCM and controls groups

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Captur, PhD, Principal Investigator — University College, London
Locations (1):
- Royal Free Hospital NHS Trust (RFH), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No